Official Title: Effect of Monazite Sands in Patients With Osteoarthritis of the Knee

Ethical committee Protocol No: 3.160.891

**Enrolment Log** 

Document date: May 2nd, 2019

## SUBJECT ENROLMENT LOG

**Study brief Title:** Effects of Sand Treatment on Osteoarthritis

Official Title: Effect of Monazite Sands in Patients with Osteoarthritis of the Knee

Ethical committee Protocol No: 3.160.891 Unique Protocol ID: T015-M02-2019AF002

| S.No. | Identifier/initials<br>if applicable | Screening Date (dd/mm/yyyy) | Exclusion met?1 | If ineligible,<br>specify reason<br>for ineligibility | Signed the inform consent? | Enrolment date (dd/mm/yyyy) | Subject ID<br>If No,<br>reasons | Investigato<br>r Initials<br>and Date |
|---|---|---|---|---|---|---|---|---|
| | | | Yes O No O | | Yes O No O | | | |
| | | | Yes O No O | | Yes O No O | | | |
| | | | Yes O No O | | Yes O No O | | | |
| | | | Yes O No O | | Yes O No O | | | |
| | | | Yes O No O | | Yes O No O | | | |
| | | | Yes O No O | | Yes O No O | | | |

<sup>&</sup>lt;sup>1</sup>Exclusion Criteria: A) History of previous knee surgery. B) History of fracture in the knee region. C) History of any secondary OA associated with any cystic arthropathy. D) Any treatment for the knee with methotrexate. E) History of hemorrhagic disorders. F) History of any infiltration of the knee during the previous 6 months (eg corticosteroids and hyaluronic acid). G) Morbid obesity. H) History of severe psychiatric disorders. I) History of skin cancer.

| Signature of the Principal Investigator: | Date: |
|-------------------------------------------|-------|
| Digitature of the filmerpul investigatory | Duce |